CLINICAL TRIAL: NCT07091214
Title: Precision Allograft Rejection Using Novel Diagnostic Approaches in Kidney Transplantation - Allograft Transcriptomics Landscape Analysis Using Sequencing (the PANDA-Kids-ATLAS Study)
Brief Title: Molecular Transcriptomics in Diagnosing Pediatric Kidney Transplant Rejection: the PANDA-Kids-ATLAS Study
Status: Not yet recruiting | Type: Observational
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Collaborators: Paris Cardiovascular Research Center (Inserm U970) (Other Government)
Responsible Party: Sponsor
Other Study IDs: Transcriptomics_PED_001
Record Dates: First submitted 2025-05-22; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Kidney Rejection Transplant
Keywords: transcriptomics; pediatric kidney transplantation; allograft rejection; precision diagnosis; molecular classifiers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Classic rejection profile: Active/chronic AMR or TCMR
- Group 2: Other rejection profiles: Probable AMR, MVI+DSA- C4d-, borderline or mixed rejection
- Group 3: Other diagnoses: CMV, CNI toxicity, recurrence, BK nephropathy
- Group 4: Normal biopsies: No lesions (normal biopsy results)

SUMMARY:
Children with kidney failure have markedly increased mortality and face repeated transplantation over their lifetime due to limited allograft half-life (12-15 years). Current biopsy-based diagnoses of rejection (using Banff 2022 criteria) suffer from variability and limited sensitivity. PANDA-Kids-ATLAS will analyze up to 600 pediatric FFPE kidney biopsies across multiple centres using the Banff Human Organ Transplant (B-HOT) NanoString panel to develop and validate molecular classifiers of AMR, TCMR and related phenotypes. A secure REDCap database will integrate molecular, pathological and clinical data, aiming to improve early detection, personalize therapy, and enhance long-term graft survival and patient quality of life.

DETAILED DESCRIPTION:
The study builds a deeply phenotyped international cohort of pediatric transplant patients (<21 years) with both retrospective (2014-present) and prospective (through Dec 2027) biopsy sampling. Four diagnostic "baskets" (classical AMR/TCMR; probable ABMR/MVI; other injury; normal) will each contribute equal numbers of cases for classifier validation (Part A) and real-world prevalence samples for outcome association (Part B). FFPE blocks will be centrally reviewed via Banff 2022 automated and expert pathologist interpretation, then processed by NanoString nCounter® using the 770-gene B-HOT panel. Stratified random sampling, robust QC, and integration with clinical/immunological parameters in REDCap will underpin molecular classifier development and validation. Follow-up includes clinical outcomes and graft function monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 21 years
* Single kidney transplant recipients (deceased or living donor)
* Written informed consent from patients/guardians

Exclusion Criteria:

* Multi-organ transplantation history
* Biopsies with insufficient tissue

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric kidney transplant recipients
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of Molecular Classifiers for Kidney Allograft Rejection Using Banff Human Organ Transplant (B-HOT) Gene Panel via NanoString nCounter® | 3 years
  Molecular signatures (molecular classifiers) will be identified through bulk transcriptomic analysis utilizing the validated Banff Human Organ Transplant (B-HOT) gene panel, consisting of 770 rejection- and tolerance-related genes. Formalin-fixed, paraffin-embedded (FFPE) biopsy samples from pediatric kidney transplant recipients will be processed and analyzed using the NanoString nCounter® platform. Specifically, molecular classifiers distinguishing classical antibody-mediated rejection (AMR), T-cell mediated rejection (TCMR), and novel Banff 2022 antibody-mediated rejection-related categories-including microvascular inflammation with donor-specific antibodies and negative C4d staining (MVI+DSA-C4d-) and probable antibody-mediated rejection (pABMR)-will be quantified and reported. Classifier results will be summarized as normalized gene expression profiles, enabling clear discrimination among different categories of rejection and non-rejection biopsies.

SECONDARY OUTCOMES:
Integration of Molecular Classifiers with Clinical Parameters into an Archetype-based Diagnostic System for Kidney Allograft Rejection | 3 years
  An archetype-based diagnostic framework will be generated by integrating transcriptomic molecular classifiers (quantified using NanoString nCounter® platform and Banff Human Organ Transplant (B-HOT) gene panel) with clinical parameters. Clinical parameters include patient demographics (age, sex), transplant characteristics, and clinical outcomes (e.g., serum creatinine, estimated glomerular filtration rate (eGFR), proteinuria, biopsy indication). The integrated diagnostic system will provide archetype-based patient profiles to enhance diagnostic precision and personalized clinical management. Aggregation will be performed using multidimensional modeling techniques (principal component analysis, cluster analyses) and classification algorithms (logistic regression, random forest), providing composite diagnostic archetypes.
  Unit of measure: Composite diagnostic archetype (multidimensional categorical profile)
Integration of Molecular Classifiers with Biological and Immunological Parameters into an Archetype-based Diagnostic System for Kidney Allograft Rejection | 3 years
  An archetype-based multidimensional diagnostic framework will be developed by combining transcriptomic molecular classifiers (from the NanoString nCounter® platform and B-HOT gene panel) with biological and immunological parameters. Specifically, this will include immunological markers such as donor-specific antibodies (DSA), C4d staining, complement factors, and inflammatory biomarkers (e.g., cytokines, chemokines, immune cell subset analysis). The integration will be conducted through bioinformatics approaches and supervised machine learning models, culminating in archetypal patient classification based on immune and biological profiles.
  Unit of measure: Composite immuno-biological archetype (multidimensional categorical profile)

OTHER OUTCOMES:
Correlation of Archetype-based Diagnostic Profiles with Kidney Allograft Clinical Outcomes | 3 years
  The correlation between archetype-based diagnostic profiles (derived from molecular, clinical, biological, and immunological data integration) and kidney allograft clinical outcomes will be assessed.
  Clinical outcomes include: 1) Incidence of acute rejection episodes (percentage [%] of patients experiencing biopsy-proven acute rejection, confirmed via Banff 2022 criteria). 2) Allograft survival rate (% graft survival, defined as a functioning graft without dialysis dependence or retransplantation). 3) Allograft function decline (rate of decline in eGFR [mL/min/1.73 m²/year], calculated from serum creatinine using the Schwartz pediatric formula).
  Each of these clinical outcomes will be individually correlated with the diagnostic archetype profiles using statistical analyses such as Kaplan-Meier survival curves, Cox proportional hazard models (for allograft survival and rejection-free survival), and regression analysis (for eGFR decline).

CONTACTS AND LOCATIONS:
Overall Officials: Evgenia Preka, MD, PhDc, Principal Investigator — INSERM U970; Alexandre Loupy, MD, PhD, Study Chair — INSERM U970; Valentin Goutaudier, MD, PhD, Study Chair — INSERM U970
Locations (1):
- Paris Institute for Transplantation and Organ Regeneration (PITOR), Paris, France

IPD SHARING:
Plan to Share IPD: Yes
molecular classifiers results
Supporting Information: Study Protocol, ICF
Time Frame: after the completion and publication of the study
Access Criteria: Participating centres' PI can contact the PI of the study for access in their center's results.
URL: https://certain-registry.kikli.uni-heidelberg.de/

REFERENCES:
- [Background] Sablik M, Sannier A, Raynaud M, Goutaudier V, Divard G, Astor BC, Weng P, Smith J, Garro R, Warady BA, Zahr RS, Twombley K, Dharnidharka VR, Dandamudi RS, Fila M, Huang E, Sellier-Leclerc AL, Tonshoff B, Rabant M, Verine J, Del Bello A, Berney T, Boyer O, Catar RA, Danger R, Giral M, Yoo D, Girardin FR, Alsadi A, Gourraud PA, Morelon E, Le Quintrec M, Try M, Villard J, Zhong W, Bestard O, Budde K, Chauveau B, Couzi L, Brouard S, Hogan J, Legendre C, Anglicheau D, Aubert O, Kamar N, Lefaucheur C, Loupy A. Microvascular Inflammation of Kidney Allografts and Clinical Outcomes. N Engl J Med. 2025 Feb 20;392(8):763-776. doi: 10.1056/NEJMoa2408835. Epub 2024 Oct 24. PMID 39450752
- [Background] Halloran PF, Madill-Thomsen KS, Bohmig G, Bromberg J, Budde K, Barner M, Mackova M, Chang J, Einecke G, Eskandary F, Gupta G, Myslak M, Viklicky O, Akalin E, Alhamad T, Anand S, Arnol M, Baliga R, Banasik M, Bingaman A, Blosser CD, Brennan D, Chamienia A, Chow K, Ciszek M, de Freitas D, Deborska-Materkowska D, Debska-Slizien A, Djamali A, Domanski L, Durlik M, Fatica R, Francis I, Fryc J, Gill J, Gill J, Glyda M, Gourishankar S, Grenda R, Gryczman M, Hruba P, Hughes P, Jittirat A, Jurekovic Z, Kamal L, Kamel M, Kant S, Kasiske B, Kojc N, Konopa J, Lan J, Mannon R, Matas A, Mazurkiewicz J, Miglinas M, Muller T, Narins S, Naumnik B, Patel A, Perkowska-Ptasinska A, Picton M, Piecha G, Poggio E, Bloudickova SR, Samaniego-Picota M, Schachtner T, Shin S, Shojai S, Sikosana MLN, Slatinska J, Smykal-Jankowiak K, Solanki A, Veceric Haler Z, Vucur K, Weir MR, Wiecek A, Wlodarczyk Z, Yang H, Zaky Z. Subthreshold rejection activity in many kidney transplants currently classified as having no rejection. Am J Transplant. 2025 Jan;25(1):72-87. doi: 10.1016/j.ajt.2024.07.034. Epub 2024 Aug 6. PMID 39117038
- [Background] Mengel M, Loupy A, Haas M, Roufosse C, Naesens M, Akalin E, Clahsen-van Groningen MC, Dagobert J, Demetris AJ, Duong van Huyen JP, Gueguen J, Issa F, Robin B, Rosales I, Von der Thusen JH, Sanchez-Fueyo A, Smith RN, Wood K, Adam B, Colvin RB. Banff 2019 Meeting Report: Molecular diagnostics in solid organ transplantation-Consensus for the Banff Human Organ Transplant (B-HOT) gene panel and open source multicenter validation. Am J Transplant. 2020 Sep;20(9):2305-2317. doi: 10.1111/ajt.16059. Epub 2020 Jun 27. PMID 32428337
- [Background] Zielinski D, Goutaudier V, Sablik M, Divard G, Aubert O, Piedrafita A, Mezine F, Dagobert J, Certain A, Robin B, Gueguen J, Rabant M, Duong van Huyen JP, Sannier A, Randoux-Lebrun C, Maanaoui M, Lionet A, Gibier JB, Gnemmi V, Le Quintrec M, Chauveau B, Vermorel A, Couzi L, Bestard O, Elias M, Louis K, Rosales IA, Smith RN, Kung VL, Anglicheau D, Legendre C, Del Bello A, Huang E, Adam B, Kamar N, Colvin RB, Mengel M, Lefaucheur C, Loupy A. Molecular diagnosis of kidney allograft rejection based on the Banff Human Organ Transplant gene panel: A multicenter international study. Am J Transplant. 2025 Aug;25(8):1631-1642. doi: 10.1016/j.ajt.2025.04.025. Epub 2025 May 8. PMID 40345499
- [Background] Fichtner A, Gauche L, Susal C, Tran TH, Waldherr R, Krupka K, Guzzo I, Carraro A, Oh J, Zirngibl M, Weitz M, Konig J, Buscher A, Berta L, Simon T, Awan A, Rusai K, Topaloglu R, Peruzzi L, Printza N, Kim JJ, Weber LT, Melk A, Pape L, Rieger S, Patry C, Hocker B, Tonshoff B; CERTAIN study group. Incidence, risk factors, management strategies, and outcomes of antibody-mediated rejection in pediatric kidney transplant recipients-a multicenter analysis of the Cooperative European Paediatric Renal Transplant Initiative (CERTAIN). Pediatr Nephrol. 2025 Feb;40(2):491-503. doi: 10.1007/s00467-024-06487-2. Epub 2024 Sep 16. PMID 39283519
- See also: CERTAIN registry protocol for participating centers via CERTAIN — https://certain-registry.kikli.uni-heidelberg.de/